CLINICAL TRIAL: NCT05926440
Title: Phase 3, Multi-center, Observer-blind, Randomized, Controlled Study to Evaluate the Immunogenicity and Safety of SCB-2023 Vaccine Administered as a Booster Dose to Adults Who Previously Received COVID-19 Vaccine
Brief Title: Immunogenicity and Safety Study of SCB-2023 Vaccine as a Booster in Adults
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: we has selected a new candidate vaccine which is monovalent.
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLO-SCB-2023-002
Record Dates: First submitted 2023-06-08; First posted 2023-07-03 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Injections, Intramuscular; SCB-2019 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCB-2023 arm (Experimental): Participants will receive one booster dose with SCB-2023 vaccine on Day 1
  Interventions: Biological: SCB-2023 vaccine (trivalent), a recombinant SARS-CoV-2 trimeric S-protein subunit vaccine for COVID-19; intramuscular injection
- SCB-2019 arm (Active Comparator): Participants will receive one booster dose with SCB-2019 vaccine on Day 1
  Interventions: Biological: SCB-2019 (monovalent), a recombinant SARS-CoV-2 trimeric S-protein subunit vaccine for COVID-19; intramuscular injection

INTERVENTIONS:
Biological: SCB-2023 vaccine (trivalent), a recombinant SARS-CoV-2 trimeric S-protein subunit vaccine for COVID-19; intramuscular injection — SCB-2023 vaccine (trivalent), a recombinant SARS-CoV-2 trimeric S-protein subunit vaccine for COVID-19; intramuscular injection
  Arms: SCB-2023 arm
Biological: SCB-2019 (monovalent), a recombinant SARS-CoV-2 trimeric S-protein subunit vaccine for COVID-19; intramuscular injection — SCB-2019 (monovalent), a recombinant SARS-CoV-2 trimeric S-protein subunit vaccine for COVID-19; intramuscular injection
  Arms: SCB-2019 arm

SUMMARY:
The purpose of this study is to assess the immunogenicity and safety of SCB-2023 trivalent vaccine compared to the prototype SCB-2019 monovalent vaccine in participants previously vaccinated with 3 doses of inactivated COVID-19 vaccine ≥6 months prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age.
* Individuals willing and able to comply with study requirements, including all scheduled visits, vaccinations, laboratory tests and other study procedures.
* Individuals willing and able to give an informed consent, prior to screening.
* Healthy participants or participants with pre-existing medical conditions who are in a stable medical condition.
* Individuals who received three doses of inactivated COVID-19 vaccine.

Exclusion Criteria:

* Body temperature >37.8°C (axillary), or any acute illness at baseline.
* Confirmed SARS-CoV-2 infectionor with known history of COVID-19.
* Individuals who have received an investigational or licensed COVID-19 vaccine prior to Day 1 (except for inactivated COVID-19 vaccine).
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy.
* Any progressive unstable or uncontrolled clinical conditions.
* Individuals who are pregnant, or breastfeeding, or planning to become pregnant while enrolled in this study or during the study period.
* History of severe adverse reaction associated with a vaccine or severe allergic reaction.
* History of malignancy within 1 year before screening.
* Individuals who have received any other investigational product.
* Individuals who have received any other licensed vaccines within 14 days prior to enrollment.
* Treatment with Rituximab or any other anti-CD20 monoclonal antibodies.
* Known bleeding disorder that would, in the opinion of the investigator, contraindicate i.m. injection.
* Administration of intravenous immunoglobulins and/or any blood products.
* Any condition that, in the opinion of the investigator, would interfere with the primary study objectives or pose additional risk to the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
To demonstrate that SCB-2023 vaccine elicits an immune response superior to SCB-2019 for Omicron BA.5 | Day 15
  GMT ratio
To demonstrate that SCB-2023 vaccine elicits an immune response superior to SCB-2019 for Omicron XBB.1.5 | Day 15
  GMT ratio
Assess the reactogenicity of SCB-2023 vaccine compared to SCB-2019 vaccine | Day 7
  Proportion of participants with local and systemic AEs
Assess the safety of SCB-2023 vaccine compared to SCB-2019 vaccine | Day 29
  Proportion of participants with unsolicited AEs
Assess the safety of SCB-2023 vaccine compared to SCB-2019 vaccine | Up to 1 year post-vaccination
  Proportion of participants with SAE, AEs leading to early termination from study, MAAEs, and AESIs

SECONDARY OUTCOMES:
Non-inferiority with respect to ratio of the geometric mean of Omicron BA.5 titer in SCB-2023 recipients and SARS-CoV-2 Delta titers in SCB-2019 recipients, as measured by virus neutralization assay. | Day 15
  GMT ratio
Geometric mean titers elicited by SCB-2023 vaccine and SCB-2019 vaccine by virus neutralization assay against Omicron BA.5 and Omicron XBB1.5. | Day 1, 15, 180
  GMTs; GMFRs; SCRs; Proportion of participants with antibody titer ≥ LLoQ
Geometric mean fold rise elicited by SCB-2023 vaccine and SCB-2019 vaccines by virus neutralization assay against Omicron BA.5 and Omicron XBB1.5 | Day 1, 15, 180
  GMFRs
Proportion of subjects with seroconversion by virus neutralization assay against Omicron BA.5 and Omicron XBB1.5 | Day 1, 15, 180
  SCRs
Proportion of subjects with antibody titer >=LLOQ by virus neutralization assay against Omicron BA.5 and Omicron XBB1.5 | Day 1, 15, 180
  Proportion of participants with antibody titer ≥ LLoQ
Geometric mean titers elicited by SCB-2023 vaccine and SCB-2019 vaccine by virus neutralization assay against SARS-CoV-2 variants of concern | Day 1, 15
  GMTs
Geometric mean fold rise elicited by SCB-2023 vaccine and SCB-2019 vaccines by virus neutralization assay against SARS-CoV-2 variants of concern | Day 1, 15
  GMFRs
Proportion of subjects with seroconversion by virus neutralization assay against SARS-CoV-2 variants of concern | Day 1, 15
  SCRs
Proportion of subjects with antibody titer >=LLOQ by virus neutralization assay against SARS-CoV-2 variants of concern | Day 1, 15
  Proportion of participants with antibody titer ≥ LLoQ

CONTACTS AND LOCATIONS:
Locations (3):
- Philippines (3):
  - Health Index Multispecialty Clinic, Manila
  - Manila Doctors Hospital, Manila
  - Tropical Disease Foundation, Putatan